CLINICAL TRIAL: NCT06647654
Title: Real World Impact and Effectiveness of ABRYSVO® Vaccination During Pregnancy Against RSV Illness in Infants
Brief Title: Impact and Effectiveness of ABRYSVO® Vaccination During Pregnancy
Acronym: BERNI
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: iTrials S.A. (Unknown)
Responsible Party: Sponsor
Other Study IDs: C3671068; NCT06647654 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Syncytial Virus; Respiratory Tract Diseases
Keywords: Vaccine; Effectiveness; Pregnancy; Maternal; Immunization; ABRYSVO; Respiratory Syncytial Virus; Lower respiratory tract disease; Infants; Hospitalized; Hospitalization; Test Negative Design; Case control; Retrospective; Cohort; Ecologic; Respiratory outcomes; Prefusion F protein-based
MeSH Terms: conditions — Respiratory Tract Diseases | interventions — abrysvo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Standard of care RSV testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cases (Test Negative Design and Cohort Design): Infants who meet the respiratory case definition and test positive for RSV (result obtained from standard of care (SOC) testing).
  Interventions: Biological: ABRYSVO
- Controls (Test Negative Design): Infants who meet the respiratory case definition and test negative for RSV (result obtained from standard of care (SOC) testing).
  Interventions: Biological: ABRYSVO
- Ecologic Cohort (Ecologic Before-and-After Design): Aggregated data on study outcomes from five historical RSV seasons and from 2024-2026 RSV seasons (data during the COVID-19 pandemic are excluded).
  Interventions: Biological: ABRYSVO

INTERVENTIONS:
Biological: ABRYSVO — Test Negative Design: This is a non-interventional retrospective study; therefore, ABSYRVO vaccine has already been administered according to the standard of care. ABRYSVO is a bivalent RSV prefusion F protein-based vaccine (RSVpreF) composed of two prefusion F proteins to protect against both RSV-A and RSV-B.
  Ecologic Before-and-After Design: This is an ecologic before-and-after study using aggregated data; as such, the 'exposure' of interest is time before ABRYSVO program implementation (i.e., five historical pre-ABRYSVO RSV seasons) and time after ABRYSVO implementation (i.e., post-ABRYSVO RSV seasons: 2024-2026).

SUMMARY:
This study will be conducted in collaboration with a research network of independent hospital sites to evaluate the vaccine effectiveness (VE) and impact of ABRYSVO vaccination during pregnancy in a real-world population over multiple seasons, which began in 2024 across Argentina and beginning in 2025 in Uruguay. We will use three retrospective design approaches in this study:

(i) a test negative design (TND) to evaluate real-world VE of maternal ABRYSVO against RSV-associated outcomes in infants;

(ii) a descriptive cohort design to evaluate the clinical evolution of infants hospitalized with RSV-positive lower respiratory tract disease (LRTD); and

(iii) an ecologic before-and-after design to evaluate the impact of ABRYSVO vaccination during pregnancy on infant RSV-associated and all-cause respiratory outcomes.

DETAILED DESCRIPTION:
This hospital-based retrospective study will be conducted in a research network of independent hospital sites. We will collect data from hospital medical records, supplemented with information from vaccine registries. This study will use three retrospective design approaches: a test negative design (TND) to evaluate real-world vaccine effectiveness (VE) of maternal ABRYSVO against RSV-associated LRTD hospitalization and other outcomes in infants, a descriptive cohort design to evaluate the clinical features of infants hospitalized with RSV-positive LRTD, and an ecologic before-and-after design to evaluate the impact of ABRYSVO vaccination during pregnancy on infant RSV-associated and all-cause respiratory outcomes.

The TND study will include infants through 9 months of age who were admitted to one of the participating hospital sites with symptoms of respiratory infection, born at 32 weeks of gestational age or greater, met the definition of LRTD, had a respiratory specimen collected with an RSV test result through standard of care testing, born 14 days or more after start of the first seasonal ABRYSVO vaccination campaign, and born to individuals who were expected to reach the indicated ABRYSVO vaccination window during a local ABRYSVO vaccination season. To complement the VE estimates generated in the TND study, we will use the cases from the primary objective of the TND analysis as a cohort of participants to describe the endpoints in the descriptive cohort study. The ecologic before-and-after study will include information for infants and children ≤24 months of age meeting eligibility criteria in post-ABRYSVO program implementation years and in several historical RSV seasons pre-ABRYSVO program implementation.

For the TND study, a multivariable logistic regression model, adjusted for confounding, will be used to compute an adjusted odds ratio (aOR), comparing the odds of maternal ABRYSVO vaccination during pregnancy between test-positive cases and test-negative controls. VE will be estimated as (1-aOR) x 100%. Secondary and exploratory objectives will evaluate VE estimates stratified by several characteristics. For the descriptive cohort study of RSV-positive LRTD hospitalized infants ≤9 months of age (i.e., the cases from the primary objective of the TND study), infant characteristics, timing, severity/clinical features, and use of healthcare resources during the index hospitalization will be described. For the ecologic before-and-after study, the impact of maternal ABRYSVO introduction on rates of RSV-associated and all-cause outcomes among infants ≤6 months (compared with older age groups) over multiple RSV seasons will be described overall and by epidemiological week, calendar year, calendar month, age group, and hospital site. These analyses will begin in the 2024 RSV season in Argentina and continue in future RSV seasons in Argentina and Uruguay (2025 and 2026), with comparison to several pre-ABRYSVO implementation seasons. Quasi-experimental approaches will also be used to quantitatively compare incidence of study outcomes among infants aged ≤6 months with older age groups.

ELIGIBILITY:
Test Negative Design Inclusion Criteria:

1. Infants ≤9 months (≤270 days) of age on the index date.
2. Index date within the time period for data collection (approximately 01 April to 30 September in 2024, 2025, or 2026).
3. Infants born at 32 weeks of gestational age or greater.
4. Hospitalized for at least 24 hours with LRTD (symptoms related to LRTD might be absent at the time of admission but if they develop within the first 24 hours of hospitalization, the criteria for LTRD will be considered met), and specimen collected for RSV within 10 days prior to hospital admission through 3 days after a hospital admission through SOC testing.
5. Infant date of birth 14 days or more after start of the first seasonal ABRYSVO vaccination campaign, to ensure potential to have been born to an ABRYSVO-vaccinated individual.
6. Infant born to individuals who were expected (based on estimated date of delivery) to reach the indicated ABRYSVO vaccination window (320/7 to 366/7 weeks' gestation) during a local ABRYSVO vaccination season.

Test Negative Design Exclusion Criteria:

1. Received any licensed or investigational RSV preventive product (e.g., Palivizumab, Nirsevimab, active RSV vaccine) since birth.
2. Received ≥1 blood transfusion or other blood products containing antibody (e.g., fresh frozen plasma) since birth.
3. Born to individual who received any other licensed or investigational RSV vaccine during pregnancy.
4. Born to individual for whom ABRYSVO vaccination status cannot be confirmed in available data sources.
5. Infants with LRTD that require hospitalization for reasons other than clinical criteria (e.g., for social reasons, other medical condition in an infant with LRTD without hospitalization criteria).

Cohort Design Inclusion Criteria:

1. RSV positive cases ≤9 months of age from the TND study.

Cohort Design Exclusion Criteria: None.

Ecologic Before-and-After Design Inclusion Criteria:

1. Infants and children ≤24 months of age on the index date.
2. Index date during the calendar years for data collection (pre- or post-ABRYSVO program implementation.
3. Meets ≥1 outcome definition during the time period for data collection.

Ecologic Before-and-After Design Exclusion Criteria: None.

Ages: 0 Years to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Test Negative Design: All infants through 9 months of age who were admitted to one of the participating hospital sites with symptoms of respiratory infection, born at 32 weeks of gestational age or greater, met the definition of LRTD, had a respiratory specimen collected with an RSV test result through standard of care testing, born 14 days or more after start of the first seasonal ABRYSVO vaccination campaign, and born to individuals who were expected to reach the indicated ABRYSVO vaccination window during a local ABRYSVO vaccination season.
  Cohort Design: RSV positive cases from the TND study.
  Ecologic Before-and-After Design: All infants and children ≤24 months of age admitted to one of the participating hospital sites and meeting eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
RSV-associated LRTD hospitalization among infants | From birth through 6 months of age
  Lab-confirmed RSV-positive LRTD hospitalization occurring ≤180 days after birth

SECONDARY OUTCOMES:
RSV-associated severe LRTD hospitalization among infants | From birth through 6 months of age
  Lab-confirmed RSV-positive severe LRTD hospitalization occurring ≤180 days after birth
RSV-associated LRTD hospitalization among infants, stratified by temporal and clinical characteristics | From birth through 6 months of age
  Lab-confirmed RSV-positive LRTD hospitalization occurring ≤180 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671068